CLINICAL TRIAL: NCT05602129
Title: A Multi-center, Randomized, Open, Positive-controlled Two-stage Phase II Clinical Study to Evaluate the Efficacy, Safety and PK/PD Profiles of Anticoagulation of HSK36273 for Injection in Continuous Renal Replacement Therapy Subjects
Brief Title: A Clinical Study to Evaluate the Efficacy, Safety and PK/PD Profiles of Anticoagulation of HSK36273 for Injection in Continuous Renal Replacement Therapy Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK36273-201
Record Dates: First submitted 2022-10-16; First posted 2022-11-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Renal Replacement Therapy
Keywords: Renal Replacement Therapy; Anticoagulants
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK36273 Continuous infusion (Experimental): Drug:HSK36273 Administration mode:Continuous infusion
  Interventions: Drug: HSK36273
- HSK36273 Bolus+Continuous infusion (Experimental): Drug:HSK36273 Administration mode:Bolus+Continuous infusion
  Interventions: Drug: HSK36273
- Heparin sodium (Active Comparator): Drug:Heparin sodium Administration mode:Bolus+Continuous infusion
  Interventions: Drug: Heparin sodium

INTERVENTIONS:
Drug: HSK36273 — HSK36273
  Arms: HSK36273 Bolus+Continuous infusion; HSK36273 Continuous infusion
Drug: Heparin sodium — Heparin sodium
  Arms: Heparin sodium

SUMMARY:
This study is divided into Stage I and Stage II. It is planned to include 156 subjects who need CRRT treatment for more than 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 and ≤80;
2. 16 kg/m2 ≤BMI≤35 kg/m2;
3. Those who need CRRT treatment for more than 48 hours and plan to use CVVHDF treatment mode for femoral vein puncture;
4. Subjects or their guardians voluntarily sign the informed consent form in writing before any procedure related to the study starts, fully understand the purpose and significance of this trial, and are willing to comply with the trial protocol.

Exclusion Criteria:

1. Those who are known to be allergic to heparin, heparin drugs, investigational drugs or non-active ingredients of study intervention;
2. Subjects with severe coagulation dysfunction or bleeding tendency three months before the screening, such as HIT (heparin-induced thrombocytopenia), ITP (idiopathic thrombocytopenia purpura), TTP (thrombocytopenia purpura), persistent systolic blood pressure>200 mmHg or diastolic blood pressure>120 mmHg, active gastrointestinal bleeding, intracranial hemorrhage, cerebral aneurysm, severe retinopathy bleeding, hemophilia, hemolytic uremic syndrome, stroke, acute coronary syndrome;
3. Those who have undergone major cardiac surgery or craniocerebral surgery within 3 months before screening and who are judged by the study doctor to be at risk of serious bleeding;
4. Those whose platelet ≤ 50*109/L and/or INR>1.8 and/or aPTT>55s at screening;
5. Those who need to combine other blood purification methods such as blood perfusion or ECMO;
6. The time from the point of randomization to the last use of anticoagulants (low-molecular-weight heparin, warfarin, apixaban, bivalirudin, etc.), antiplatelet drugs (clopidogrel, aspirin, etc.), fibrinolytic drugs (urokinase, etc.) is shorter than the 5 half-lives of the drug or the duration of drug efficacy (calculated by the longest time);
7. The time of administration is shorter than 1 half-life of low-molecular-weight heparin from the last preventive dose;
8. Child-Pugh liver function is grade C in screening period;
9. Those with positive hepatitis C antibody or HIV antibody screening;
10. Pregnant and lactating women; women or men with fertility are unwilling to use contraception throughout the study period; subjects with pregnancy plans within 6 months after the study (including male subjects);
11. Those who have participated in clinical trials of other drugs within 3 months before screening (defined as having received investigational drug or placebo);
12. Other conditions that the investigator judges are not suitable for the subject to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Filter life | Day1 to Day5
  the time from the start of administration to the first filter replacement and the average filter using time during the treatment period
Times of filter replacement | Day1 to Day5
  the times of filter replacement within 120h after starting administration
Coagulation grade of filter and pipeline | Day1 to Day5
  Clotting in the dialyser and the air traps as evaluated by a scale from 0 to 3

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No